CLINICAL TRIAL: NCT01760980
Title: Pivotal Bioequivalence Study of Exemestane 25 mg Tablets Under Fasting Conditions in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development halted by management
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PXL209003
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Rate and extend of absorption of Exemestane
MeSH Terms: interventions — exemestane

ARMS (2):
- Test product (B) (Experimental): B: Subjects receive Exemestane 25 mg tablets under fasting conditions
  Interventions: Drug: Test product (B) Exemestane
- Reference product (A) (Active Comparator): A: Subjects receive Aromasin 25 mg tablets on two occasions under fasting conditions
  Interventions: Drug: Reference product (A) Aromasin (Exemestane)

INTERVENTIONS:
Drug: Reference product (A) Aromasin (Exemestane) — Aromasin tablets will be administered under fasting conditions on two occasions
  Other Names: Aromasin (Exemestane) 25 mg tablets
  Arms: Reference product (A)
Drug: Test product (B) Exemestane — Exemestane tablets will be administered under fasting conditions on one occasion
  Other Names: Exemestane 25 mg tablets
  Arms: Test product (B)

SUMMARY:
The objective of this study is to assess the bioequivalence of the test product, Exemestane 25 mg tablets of Actavis Group PTC ehf. Iceland, and the reference product, Aromasin® (exemestane) 25 mg tablets of Pharmacia & Upjohn Company, Division of Pfizer Inc., New York, United States of America in healthy male and postmenopausal female subjects, under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, 18 to 55 years of age and postmenopausal female subjects, 18 years to not older than 75 years of age (inclusive at time of screening).
2. Body Mass Index (BMI) between 19 and 33 kg/m2 (relates to a body mass within 15% of ideal body mass for height and age).
3. Body mass not less than 50 kg.
4. Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
5. Non-smoker or mild to moderate smoker (≤ 10 cigarettes daily).
6. Females, if:

   * Serum follicle-stimulating hormone (FSH) ≥ 25.8 mIU/mL AND a serum estradiol level of ≤ 54.7 pg/mL at screening.
   * Not of childbearing potential, e.g., has been surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal.

   Note: In postmenopausal women, the value of the serum pregnancy test may be slightly increased, but if not increasing upon repeat, the female will be included in the study.

   • Not on thyroid hormone replacement therapy or on stable thyroid hormone replacement therapy for at least 3 months before the first administration of IMP.

   Not on statin therapy or on stable statin therapy for at least 3 months before the first administration of IMP.

   • Blood pressure measurements are within the acceptable ranges; or, if diagnosed with hypertension, are on stable therapy for at least 3 months before the first administration of IMP.

   Note: Treatment with calcium channel blockers is NOT allowed.
7. Written consent given for participation in the study. -

Exclusion Criteria:

1. Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
2. Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females.
3. History of regular exposure to substances of abuse (other than alcohol) within the past year.
4. Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks prior to the first administration of IMP, except for medication allowed per inclusion criteria (Section 7.3.1) or if the medication will not affect the outcome of the study in the opinion of the investigator.
5. Female hormone replacement therapy (or other medicine containing estrogen, including health food products for menopausal symptoms, as these may contain natural estrogens), within 2 weeks prior to the first administration of IMP.
6. Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks before the first administration of IMP in this study.
7. Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
8. Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
9. A major illness during the 3 months before commencement of the screening period.
10. History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
11. History of bronchial asthma or any other bronchospastic disease within the past 5 years.
12. History of epilepsy.
13. History of porphyria.
14. Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
15. Systolic blood pressure > 150 mmHg or < 95 mmHg, and/or diastolic blood pressure > 95 mmHg or < 50 mmHg in either the supine or standing position at screening.
16. Resting pulse of > 100 beats per minute or < 45 beats per minute in either the supine or standing position at screening.
17. Positive serology testing for human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C or syphilis.
18. Positive urine screen for drugs of abuse.
19. Positive pregnancy test.
20. Female subjects of premenopausal endocrine status, including pregnant and lactating women.
21. Clinically diagnosed peptic ulceration within the past 5 years.
22. History of bleeding disorders.
23. Vegetarian or any abnormal diet (for whatever reason).
24. Any specific investigational product safety concern. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
AUCt, AUCinf and Cmax of Exemestane 25 mg tablets | 0, 0.333, 0.500, 0.750, 1.000, 1.250, 1.500, 1.750, 2.000, 2.500, 3.000, 3.500, 4.000, 6.000, 8.000, 12.000, 24.000, 36.000, 48.000, 72.000 and 96.000 hours post does

CONTACTS AND LOCATIONS:
Locations (1):
- Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa), Bloemfontein, South Africa